CLINICAL TRIAL: NCT07137299
Title: POPQ Associated With Total Laparoscopic Hysterectomy - Multicenter Prospective Observational Study - POP-LAP STUDY
Brief Title: POPQ Associated With Total Laparoscopic Hysterectomy
Acronym: POP-LAP
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Silesia (Other)
Collaborators: St. Boniface Hospital (Other); Klinika Ginekologii i Ginekologii Onkologicznej CMKP (Unknown); I Klinika Położnictwa i Ginekologii, Wydział Lekarski Warszawski Uniwersytet Medyczny (Unknown)
Responsible Party: Principal Investigator, Krzysztof Nowosielski, Prof., Medical University of Silesia
Other Study IDs: POP-LAP1
Record Dates: First submitted 2025-08-02; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Uterine Fibroids (UF); Abnormal Uterine Bleeding Unrelated to Menstrual Cycle; Endometrial Hyperplasia; Pelvic Organ Prolapse (POP)
Keywords: Hysterectomy; Vaginal hysterectomy; Laparotomy; Laparoscopy; Robotic surgery; pelvic organ prolapse
MeSH Terms: conditions — Leiomyoma; Endometrial Hyperplasia; Pelvic Organ Prolapse | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Lap-hyst: Women who underwent laparoscopic hysterectomy for benign conditions
  Interventions: Other: Questionnaire and Physical Exam
- Robot-hyst: Women who underwent robotic hysterectomy for benign conditions
  Interventions: Other: Questionnaire and Physical Exam
- Vaginal-Hyst: Women who underwent vaginal hysterectomy for benign conditions
  Interventions: Other: Questionnaire and Physical Exam
- Abdom-Hyst: Women who underwent abdominal hysterectomy for benign conditions
  Interventions: Other: Questionnaire and Physical Exam
- SAH: Women who underwent supracervical abdominal hysterectomy for benign conditions
  Interventions: Other: Questionnaire and Physical Exam
- LASH: Women who underwent Laparoscopic Assisted Supracervical Hysterectomy for benign conditions
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — All study participants will be evaluated to assess:
  * Healing of the vaginal stump in the case of a total hysterectomy (normal/abnormal),
  * Symptoms of stress urinary incontinence (Ingelmann-Sundber scale, where 0 - no symptoms, Grade I - symptoms with coughing, pressure on the suprapubic area, laughing, or strenuous exertion, Grade II - loss of urine when levering, running, or climbing stairs, Grade III - loss of urine when lying down or standing without physical exertion)
  * Symptoms of an overactive bladder - present, absent
  * Symptoms of prolapse in the anterior and posterior compartments (assessed based on the POPQ scale) with an assessment of the defect site based on the de Lancey classification The examination will be performed by or with the assistance of a specialist in obstetrics and gynecology

SUMMARY:
The goal of this observational study is to evaluate the impact of different hysterectomy (removal of the uterus) techniques on the risk of pelvic organ prolapse (situation when one or more of your pelvic organs like your bladder, uterus, or rectum have dropped down or slipped out of their normal position, sometimes even bulging into the vagina) and urinary incontinence (leaking urine unexpectedly) in women aged 18-85 who underwent hysterectomy or supracervical hysterectomy (removing of the uterus without its cervix) for benign (not cancer) conditions.

The main question is: to check how different surgical technique (laparoscopic, with opening the abdomen, vaginal and robotic) increase the risk of pelvic organ prolapse or urinary incontinence There is no randomization or control group; comparisons will be made between surgery types based on clinical and questionnaire data.

Participants will:

* Receive an invitation to participate if they underwent hysterectomy between 2021-2025.
* Fill out validated quality of life questionnaires (P-QOL, POPDI-6, PFIQ-7) every two years.
* Attend follow-up clinical pelvic exams every two years to assess vaginal cuff healing, pelvic organ prolapses (POP-Q system), and urinary symptoms.

This prospective, non-commercial, multicenter study plans to enroll 2,000 women and will run from July 1, 2025, to July 1, 2036

DETAILED DESCRIPTION:
What Is This Study About? This is a long-term observational study that aims to understand whether different surgical techniques for removing the uterus affect women's risk of developing pelvic floor disorders, such as pelvic organ prolapse (POP) or urinary incontinence, after surgery.

Pelvic organ prolapse occurs when pelvic organs like the uterus or bladder drop from their normal position and push against the vaginal walls. It is a common condition, especially in women after menopause, and can significantly affect quality of life.

Why Is This Study Important? Each year, thousands of women undergo hysterectomies (surgical removal of the uterus) for non-cancerous reasons. However, it's still unclear whether certain types of hysterectomy procedures may lead to a higher or lower risk of pelvic floor problems in the years following surgery. This study seeks to provide reliable answers to help improve patient safety and long-term outcomes.

What Questions Is the Study Trying to Answer?

The main questions it aims to answer are:

* Does total laparoscopic hysterectomy increase the risk of pelvic organ prolapse or urinary incontinence compared to supracervical hysterectomy?
* Does total laparoscopic hysterectomy increase the risk of pelvic floor dysfunction compared to abdominal or vaginal approaches?
* Does the use of robotic techniques reduce the risk of pelvic floor dysfunction compared to conventional laparoscopic hysterectomy?
* Does robotic supracervical hysterectomy reduce the risk of pelvic floor dysfunction compared to standard laparoscopic supracervical hysterectomy?

Who Can Participate? The study will include about 2,000 women who had their uterus removed or partially removed between 2021 and 2025 for benign conditions.

Participants must be:

* 18 to 85 years old
* Willing to give informed consent
* Not suffering from severe chronic illness (ECOG ≥ 2)
* Not previously diagnosed with pelvic floor problems before surgery What Will Participants Be Asked to Do?

Participants will:

* Receive a letter inviting them to join the study
* Complete quality-of-life questionnaires (Prolapse Quality of Life Questionnaire (P-QOL), Pelvic Organ Prolapse Inventory 6 (POPDI-6), Pelvic Floor Impact Questionnaire short form ( PFIQ-7).every two years about symptoms related to pelvic floor dysfunction and urinary incontinence
* Undergo a gynecological exam every two years to assess healing and signs of prolapse using a standardized method (POP-Q) If a participant chooses not to have a physical exam, only questionnaire data will be used.

Where Is the Study Taking Place?

The study is being conducted at multiple leading medical centers in Poland:

* Department of Gynecology, Obstetrics and Gynecological Oncology, University Clinical Center of the Medical University of Silesia in Katowice
* Department of Gynecology and Gynecological Oncology, CMKP, Warsaw
* Department of Gynecology and Obstetrics, Medical University of Warsaw
* Department of Obstetrics and Gynecology, Szpital Zakonu Bonifratrów pw. Aniołów Stróżów w Katowice

Is the Study Safe? Yes. This is an observational study, which means no new treatments or procedures are being tested. It involves only questionnaires and routine medical exams, so there is no additional risk to the participants.

When Will the Study Take Place?

* Start date: July 1, 2025
* End date: July 1, 2036 This long observation period allows researchers to understand how pelvic floor health changes years after surgery.

What Do Researchers Hope to Achieve? The ultimate goal is to guide medical professionals and patients in choosing the most appropriate surgical technique for removing the uterus for benign causes, based on long-term outcomes. By identifying which methods are safer for pelvic floor health, this research could help reduce the number of women who develop prolapse or incontinence after surgery.

ELIGIBILITY:
Inclusion Criteria:

* persons who underwent total or subtotal hysterectomy for benign conditions regardless of the type of surgery
* agree to participate and to follow-up

Exclusion Criteria:

* having uterus
* health state - ECOG >2
* pelvic organ prolapse prior to the surgery
* surgery due to malignant conditions (ovarian, cervical or endometrial cancer)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women operated in selected time-frame in study centers for benign conditions
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2036-07-01 (Estimated); Study Completion 2037-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of different types of hysterectomy/uterine amputation on the incidence of urinary incontinence | At baseline and at 2-year intervals (Year 2, Year 4, Year 6, Year 8, and Year 10) through study completion; on average of 10 years.
  Ingelmann-Sundberg scale for symptoms of stress urinary incontinence. The Ingelmann-Sundberg scale is a grading system used to assess the severity of stress urinary incontinence (SUI). It categorizes SUI based on the degree of physical activity that provokes urine leakage. The scale has three grades, with Grade I being the mildest and Grade III the most severe.
  Grade I - Urine leakage occurs with a relevant increase in abdominal pressure, such as during coughing, sneezing, or laughing.
  Grade II - Urine leakage occurs with a lesser increase in abdominal pressure, such as during activities like running, picking up objects from the floor, or walking.
  Grade III - Urine leakage occurs with minimal physical exertion, such as during walking, stair climbing, or even while standing or lying down.
  The assessment is based on medical interview with the patient performed during clinical visit.
Assessment of the impact of different types of hysterectomy/uterine amputation on the incidence of overactive bladder. | At baseline and at 2-year intervals (Year 2, Year 4, Year 6, Year 8, and Year 10) through study completion; on average of 10 years.
  OABSS Overactive Bladder Symptom Score (OABSS) was used to assess symptoms of overactive bladder. The scale consists of 7 questions on a five-point Likert scale that refer to every symptom of OAB: 1 for nocturia, 1 for urinary frequency, 3 for urgency, 1 for urge incontinence, and 1 generic question about bladder control. The total result is scored from 0 to 28, with patients with higher scores reporting worse symptoms.
Assessment of the impact of different types of hysterectomy/uterine amputation on the incidence of pelvic organ prolapse | At baseline and at 2-year intervals (Year 2, Year 4, Year 6, Year 8, and Year 10) through study completion; on average of 10 years.
  POPQ - Pelvic Organ Prolapse-Quantification. The assessment is based on gynecological examination. The system measures the position of the most distal portion of the prolapse to the hymen level. 5 stages are described:
  * Stage 0: No prolapse
  * Stage I: Most distal prolapse is more than 1 cm above the hymen
  * Stage II: Most distal prolapse is between 1 cm above and 1 cm below the hymen
  * Stage III: Most distal prolapse is more than 1 cm below hymen but 2 cm shorter than total vaginal length
  * Stage IV: Complete eversion

SECONDARY OUTCOMES:
Complications | up to 30 days postoperatively
  Assessment of complications after hysterectomy/uterine amputation based on Clavien-Dindo Classification. The Clavien-Dindo Classification consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). It assesses the complications of the surgery in order to rank them in an objective and reproducible manner.
  Grade I - Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Grade II- Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
  Grade III - Requiring surgical, endoscopic or radiological intervention Grade IV - Life-threatening complication (including CNS complications) requiring Intensive Care Unit management Grade V - Death of a patient
Assessment of the impact of different types of hysterectomy/uterine amputation on quality of life - by using P-QOL | At baseline and at 2-year intervals (Year 2, Year 4, Year 6, Year 8, and Year 10) through study completion; on average of 10 years.
  P-QOL - Prolapse Quality of Life Questionnaire. The scale consisted of 38 questions, with 20 questions representing nine quality of life domains (general health perception, prolapse impact, role and physical limitations, social limitations, personal relationships, emotional problems, sleep/energy disturbances and symptoms severity) and 18 questions about prolapse symptoms. The responses ranged from "none/not at all" through "slightly/a little" and "moderately" to "a lot". A four-point scoring system for each item is used for severity measurement of urogenital prolapse symptoms. The questionnaire does not form the combined score. If a woman has only one domain affected and another woman has all domains affected, both will be considered symptomatic but in different aspects of life quality. Higher scores indicate a greater impairment of quality of life, and lower scores indicate a good quality of life.
Assessment of the impact of different types of hysterectomy/uterine amputation on quality of life - by using POPDI-6 | At baseline and at 2-year intervals (Year 2, Year 4, Year 6, Year 8, and Year 10) through study completion; on average of 10 years.
  POPDI-6 - Pelvic Organ Prolapse Inventory 6. The scale is a six-item questionnaire used to assess the level of distress caused by pelvic organ prolapse symptom. Each of the six items is scored on a scale, ranging from 0 to 4, where 0 represents no distress and higher scores indicate greater distress. The scores range from 0 to 24, where higher scores indicate greater distress from pelvic organ prolapse symptoms
Assessment of the impact of different types of hysterectomy/uterine amputation on quality of life - by using PFIQ-7 | At baseline and at 2-year intervals (Year 2, Year 4, Year 6, Year 8, and Year 10) through study completion; on average of 10 years.
  PFIQ-7 - Pelvic Floor Impact Questionnaire short form is a 7-item questionnaire used to assess the impact of pelvic floor disorders on a woman's quality of life. It measures the impact of urinary symptoms (UIQ-7), pelvic organ prolapse symptoms (PIPQ-7) and colorectal/anal symptoms (CRAIQ-7) on daily life. Each item is scored on a Likert scale (0, Not at all; 1, somewhat; 2, moderately; 3, quite a bit), and scores from each scale can be combined to provide an overall impact score. The score for subscale ranges from 0 to 100 and for total score - 0-300. Higher scores represent greater impact on daily life.

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Department of Gynaecology, Obstetrics and Gynaecological Oncology, University Clinical Centre, Medical University of Silesia, Katowice, Silesian Voivodeship
  - Department of Obstetrics and Gynecology, Szpital Zakonu Bonifratrów pw. Aniołów Stróżów, Katowice
  - Department of Gynecology and Obstetrics, Medical University of Warsaw, Warsaw
  - Department of Gynecology and Obstetrics, Szpital Bielański, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data (all) will be shared on request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01.07.2026 - indefinitely
Access Criteria: All academic researches on request